CLINICAL TRIAL: NCT04652739
Title: Evaluation of Lycopene in the Treatment of Erosive Oral Lichen Planus (A Randomized Clinical Trial)
Brief Title: Evaluation of Lycopene in the Treatment of Erosive Oral Lichen Planus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lycopene and lichen planus
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Erosive Lichen Planus
MeSH Terms: interventions — Prednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lycopene (Experimental)
  Interventions: Drug: Lycopene Softgel, 10 Mg
- Corticosteroids (Active Comparator)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Lycopene Softgel, 10 Mg — Patients were given 10 mg of lycopene softgel capsules once daily for two months. The active ingredient in each capsule consists of 10 mg lycopene from natural tomato extract.
  Arms: Lycopene
Drug: Prednisolone — Patients were given 40 mg of prednisolone tablets once daily in the morning for one month, afterwards, the dose was tapered along the following month. Incremental reduction of 10 mg each week for the first three weeks, followed by 5 mg reduction in the last week, was the tapering protocol in this study. The active ingredient in each tablet consists of Prednisolone metasulfobenzoate sodium 31.44 mg (equivalent to 20 mg of Prednisolone).
  Other Names: Corticosteroids
  Arms: Corticosteroids

SUMMARY:
The aim of this study was to evaluate the effect of oral lycopene and systemic steroids in the treatment of erosive oral lichen planus and compare between the two therapeutic modalities.

DETAILED DESCRIPTION:
Twenty erosive lichen planus patients were recruited and randomly assigned in one of two groups, the test (lycopene) and control (corticosteroids) group.

ELIGIBILITY:
Inclusion Criteria:

* Erosive oral lichen planus patients with severe and extensive painful erythematous, erosive and/ or ulcerative lesions who are in need for systemic corticosteroid therapy

Exclusion Criteria:

* Pregnant females and smokers.
* Patients suggestive of having lichenoid contact/drug reactions.
* Patients suffering from any systemic disease as diabetes, liver disease, renal disease, any other autoimmune or collagen disease.
* Lesions showing histological features of dysplasia.
* Patients with skin lichen planus lesions.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Pain assessment was conducted using Visual Analogue Scale (VAS) | up to 5 months
  Patients were instructed to mark a 10 cm line at a point equivalent to their present pain. The score was determined by measuring the distance in mm on the line from the "no pain" anchor to the patient's mark, providing a range of scores from 0-100. A Pain-free experience was scored zero, while the worst pain was scored 100.
Lesion size assessment | up to 5 months
  Assessment of OLP lesions was performed using the Thongprasom et al. scoring index where:
  * Score 0: No lesion/Normal mucosa.
  * Score 1: Mild white striae only.
  * Score 2: White striae with erythematous area <1cm².
  * Score 3: White striae with erythematous area >1cm².
  * Score 4: White striae with erosive area <1cm².
  * Score 5: White striae with erosive area >1cm².
  * Scores from different oral sites were added to give a final score for every patient from 0-50.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa A Bedeir, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Azza M Zaki, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Sabah A Mahmoud, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Thongprasom K, Luangjarmekorn L, Sererat T, Taweesap W. Relative efficacy of fluocinolone acetonide compared with triamcinolone acetonide in treatment of oral lichen planus. J Oral Pathol Med. 1992 Nov;21(10):456-8. doi: 10.1111/j.1600-0714.1992.tb00974.x. PMID 1460584
- [Background] Gobbo M, Rupel K, Zoi V, Perinetti G, Ottaviani G, Di Lenarda R, Bevilacqua L, Woo SB, Biasotto M. Scoring systems for Oral Lichen Planus used by differently experienced raters. Med Oral Patol Oral Cir Bucal. 2017 Sep 1;22(5):e562-e571. doi: 10.4317/medoral.21833. PMID 28809373